CLINICAL TRIAL: NCT05724628
Title: A Pilot Randomized Trial of Non-operative Versus Operative Management of Acute Appendicitis in Vulnerable Patient Populations
Brief Title: Non-operative vs. Operative Management of Acute Appendicitis in Vulnerable Patient Populations
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Project did not receive final IRB approvals. PI decided to withdrawn research study.
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Sneha Bhat, ASSISTANT PROFESSOR - Surgery, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STU-2021-0035
Record Dates: First submitted 2022-12-18; First posted 2023-02-13 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: Acute Appendicitis
MeSH Terms: conditions — Appendicitis | interventions — Anti-Bacterial Agents

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Operative Arm (Experimental): Operation (laparoscopic appendectomy) will be performed to remove appendix.
  Interventions: Procedure: Laparoscopic appendectomy
- Non-Operative Arm (Experimental): No operation will be performed, and instead, will receive intra-venous (IV) antibiotics, transitioned to by mouth (oral) antibiotics
  Interventions: Drug: Antibiotics (IV transitioned to oral)

INTERVENTIONS:
Procedure: Laparoscopic appendectomy — Subjects will receive surgery (using 3 port Laparoscopic appendectomy) to remove appendix
  Arms: Operative Arm
Drug: Antibiotics (IV transitioned to oral) — Subjects will be admitted to the hospital for antibiotic treatment, initially with IV antibiotics and then transitioned to by mouth (PO) antibiotics for the rest of the course.
  Drugs used would be anything from: zosyn, ciprofloxacin or ceftriaxone and flagyl, augmentin
  Arms: Non-Operative Arm

SUMMARY:
The overall project goal is to conduct a pilot randomized clinical trial of operative (laparoscopic appendectomy) vs nonoperative (antibiotic) management of uncomplicated acute appendicitis for vulnerable populations. Specifically, the elderly, non-English speakers, and those with economic vulnerability (low socioeconomic status and/or manual labor jobs without a non-weight lifting aspect), are three vulnerable population subsets identified. This pilot trial will provide critical preliminary data for planning and conducting a larger multi-site randomized trial.

DETAILED DESCRIPTION:
The study would involve consented subjects, once confirmed eligible to proceed after screening, will be randomly assigned to two arms:

* Group 1 - Operative Group - Operation will be performed to remove appendix.
* Group 2 - Non-operative group - No operation will be performed, and instead the subject will receive intra-venous (IV) antibiotics, transitioned to by mouth (oral) antibiotics, for treatment of appendicitis.

Aside from the routine hospital care, participants will be asked to fill out a survey for cognitive function (CAM Assessment Form), pain (Visual Analog Scale), and quality of life at the start and end of participant's hospital stay, 1-2 weeks after discharge, and again at 6 weeks after discharge from the initial hospital visit.

Participants will also be asked to participate in a qualitative interview, either by virtual visit, site visit, or phone call, at 1-2 weeks and again at about 6 weeks after discharge from the hospital. Each interview will be approximately 20-30 minutes of the participant's time.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Able to consent for the study
* Diagnosis of acute appendicitis confirmed by CT imaging

Exclusion Criteria:

* Appendicolith/fecalith on imaging
* Chronic or recurrent appendicitis
* Having received prior antibiotic treatment for other reasons within 5 days prior to study enrollment
* Hemodynamically abnormal (SBP<90 mmHg, Heart Rate (HR) >120, mmHg, Partial Pressure of Oxygen in Arterial Blood (PaO2<60), or potential of Hydrogen (pH<7.3)).
* Inability to tolerate general anesthesia (determined by surgery and anesthesiology teams)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-10 (Estimated); Primary Completion 2023-11 (Estimated); Study Completion 2023-11 (Estimated)

PRIMARY OUTCOMES:
Feasibility of the intervention as measured by the proportion of enrolled participants retained in this study | 12 months post treatment
  Feasibility of the intervention is measured by the proportion of enrolled participants who are randomized and retained in this study
Feasibility of the intervention as measured by the number of complications or adverse events | 12 months post treatment
  Feasibility of the intervention is measured by the number of complications or adverse events encountered by participants while enrolled in this study

SECONDARY OUTCOMES:
Feasibility of the intervention as measured by total length of hospital stay (Antibiotics Group) | the day of discharge (approx. 1-3 days post treatment)
  Feasibility of the intervention is measured by total number of days in inpatient hospital stay for the IV antibiotics group post treatment
Feasibility of the intervention as measured by total length of hospital stay (Operative Group) | the day of discharge (approx. 0-2 days post treatment)
  Feasibility of the intervention is measured by total number of days in inpatient hospital stay for the Operative group post laparoscopic appendectomy
Feasibility of the intervention as measured by the number of hospital readmissions or emergency room visits | 1-2 weeks post-discharge
  Feasibility of the intervention is measured by the count of the number of hospital readmissions or emergency room visits by the participants at 1-2 weeks post-discharge
Feasibility of the intervention as measured by the number of hospital readmissions or emergency room visits | 6 weeks post-discharge
  Feasibility of the intervention is measured by the count of the number of hospital readmissions or emergency room visits by the participants at 6 weeks post-discharge
Feasibility of the intervention as measured by QoL surveys | prior to discharge home (approx. 4-6 hours post treatment)
  Feasibility of the intervention is measured by administering Quality of Life (QoL) surveys using Quality of Recovery-40 questionnaire. This is a self-rated questionnaire for early postoperative quality of recovery and health status of patients. Possible scores range from 1 to 5, where higher scores indicate better quality of life (i.e., 1 = very poor and 5 = excellent)
Feasibility of the intervention as measured by QoL surveys | 1-2 weeks post-discharge
  Feasibility of the intervention is measured by administering Quality of Life (QoL) surveys using Quality of Recovery-40 questionnaire. This is a self-rated questionnaire for early postoperative quality of recovery and health status of patients. Possible scores range from 1 to 5, where higher scores indicate better quality of life (i.e., 1 = very poor and 5 = excellent)
Feasibility of the intervention as measured by QoL surveys | 6 weeks post-discharge
  Feasibility of the intervention is measured by administering Quality of Life (QoL) surveys using Quality of Recovery-40 questionnaire. This is a self-rated questionnaire for early postoperative quality of recovery and health status of patients. Possible scores range from 1 to 5, where higher scores indicate better quality of life (i.e., 1 = very poor and 5 = excellent)
Change in pain score from baseline as measured by visual analog pain scale at prior to discharge home (approx. 4-6 hours post treatment) | Baseline, prior to discharge home (approx. 4-6 hours post treatment)
  Change in pain score from baseline is measured by visual analog pain scale at prior to discharge home (approx. 4-6 hours post treatment). Possible scores range from 0-10, where 0= no pain and 10= worst pain.
Change in pain score from baseline as measured by visual analog pain scale at 1-2 weeks post discharge | Baseline, 1-2 weeks post discharge
  Change in pain score from baseline is measured by visual analog pain scale at weeks post discharge. Possible scores range from 0-10, where 0= no pain and 10= worst pain.
Change in pain score from baseline as measured by visual analog pain scale at 6 weeks post discharge | Baseline, 6 weeks post discharge
  Change in pain score from baseline is measured by visual analog pain scale at 6 weeks post discharge. Possible scores range from 0-10, where 0= no pain and 10= worst pain.
Change in cognitive function as measured by CAM assessment form at 1-2 weeks post discharge | Baseline, 1-2 weeks post discharge
  Change in cognitive function is measured by Short Confusion Assessment Method (CAM) Questionnaire at 1-2 weeks post discharge. If Inattention and at least one other item ( regarding acute change in mental status; inattention) in Box 1 of the questionnaire are checked and at least one item (regarding disorganized thinking; altered level of consciousness) in Box 2 of the questionnaire is checked, then a diagnosis of delirium is suggested.
Change in cognitive function as measured by CAM assessment form at 6 weeks post discharge | Baseline, 6 weeks post discharge
  Change in cognitive function is measured by Short Confusion Assessment Method (CAM) Questionnaire at 6 weeks post discharge. If Inattention and at least one other item ( regarding acute change in mental status; inattention) in Box 1 of the questionnaire are checked and at least one item (regarding disorganized thinking; altered level of consciousness) in Box 2 of the questionnaire is checked, then a diagnosis of delirium is suggested.
Feasibility of the intervention as measured by physical function using FRAIL scale | Baseline
  Feasibility of the intervention is measured by physical function using FRAIL scale. The Fatigue Resistance Ambulation Illness and Loss of weight (FRAIL) scale includes 5 components: Fatigue, Resistance, Ambulation, Illness, and Loss of weight. Frail scale scores range from 0-5 (i.e., 1 point for each component; 0=best to 5=worst) and represent frail (3-5), pre-frail (1-2), and robust (0) health status.
Feasibility of the intervention as measured by hospital costs for each enrolled participant (Antibiotics Group) | the day of discharge (approx. 1-3 days post treatment)
  Feasibility of the intervention is measured by accessing billing codes/hospital costs for each enrolled subject from the time they are admitted until they are discharged from the hospital.
Feasibility of the intervention as measured by hospital costs for each enrolled participant (Operative Group) | the day of discharge (approx. 0-2 days post treatment)
  Feasibility of the intervention is measured by accessing billing codes/hospital costs for each enrolled subject from the time they are admitted until they are discharged from the hospital.

CONTACTS AND LOCATIONS:
Overall Officials: Sneha Bhat, Principal Investigator — University of Texas Southwestern Medical Center

IPD SHARING:
Plan to Share IPD: No